CLINICAL TRIAL: NCT02235740
Title: An Open Label, Two-part, Phase I/Randomized Phase II Study in Subjects With Relapsed/Refractory Multiple Myeloma to Determine a Dose of Afuresertib for Administration in Combination With Carfilzomib (Part 1) and to Investigate the Safety, Pharmacokinetics, and Clinical Activity of the Combination of Afuresertib With Carfilzomib Compared With Carfilzomib Alone (Part 2)
Brief Title: A Study Conducted in Subjects With Relapsed/Refractory Multiple Myeloma (MM); to Determine Dose of Afuresertib in Combination With Carfilzomib (Part 1) and to Investigate the Safety, Pharmacokinetic and Clinical Activity of the Combination Compared With Carfilzomib Alone (Part 2)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200623
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: Open label; carfilzomib; Phase I; clinical activity; pharmacokinetics; afuresertib; relapsed; refractory; safety; multiple myeloma
MeSH Terms: conditions — Neoplasms; Recurrence; Multiple Myeloma | interventions — afuresertib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Afuresertib 125 mg+ Carfilzomib (Part 1) (Experimental): Approximately 8 subjects will receive Afuresertib 125 mg daily starting Cycle 1 Day 2 + Carfilzomib 20 mg/m^2: Cycle 1, Day 1, 2; Cycle 2, Day 1. Carfilzomib 27 mg (increased dosage of 27 mg/meter (m)^2 will be administered only if tolerated): Cycle 1, Days 8, 9, 15, and 16; Cycle 2, Days 2, 8, 9, 15, and 16; Cycle 3 and onwards, Days 1, 2, 8, 9, 15, and 16 of each cycle
  Interventions: Drug: Afuresertib; Drug: Carfilzomib
- Afuresertib 150 mg+ Carfilzomib (Part 1) (Experimental): Approximately 8 subjects will receive oral Afuresertib 150 mg daily starting Cycle 1 Day 2 + Carfilzomib 20 mg/m^2: on Cycle 1, Day 1, 2; Cycle 2, Day 1. Carfilzomib 27 mg/m^2 (increased dosage of 27 mg/m^2 will be administered only if tolerated): Cycle 1, Days 8, 9, 15, and 16; Cycle 2, Days 2, 8, 9, 15, and 16; Cycle 3 and onwards, Days 1, 2, 8, 9, 15, and 16 of each cycle
  Interventions: Drug: Afuresertib; Drug: Carfilzomib
- Afuresertib 100 mg+ Carfilzomib (Part 1) (Experimental): An additional arm with 100 mg of afuresertib may be evaluated if the other 2 arms are not tolerated. Approximately 8 subjects will receive Afuresertib 100 mg daily starting Cycle 1 Day 2 + Carfilzomib 20 mg/m^2: on Cycle 1, Day 1, 2; Cycle 2, Day 1. Carfilzomib 27 mg/m^2 (increased dosage of 27 mg/m^2 will be administered only if tolerated): Cycle 1, Days 8, 9, 15, and 16; Cycle 2, Days 2, 8, 9, 15, and 16; Cycle 3 and onwards, Days 1, 2, 8, 9, 15, and 16 of each cycle
  Interventions: Drug: Afuresertib; Drug: Carfilzomib
- Afuresertib/carfilzomib (Part 2) (Experimental): Approximately 50 subjects will receive Afuresertib Recommended Phase 2 Dose (RP2D) daily starting Cycle 1 Day 1 + Carfilzomib 20 mg/m^2 Cycle 1, Day 1, 2. Carfilzomib 27 mg (increased dosage of 27 mg/m^2 will be administered only if tolerated): Cycle 1, Days 8, 9, 15 and 16; Cycle Days 1, 2, 8, 9, 15 and 16 of each cycle; Cycle 3 and onwards, Days 1, 2, 8, 9 and 15 and 16 of each cycle.
  Interventions: Drug: Afuresertib; Drug: Carfilzomib
- Carfilzomib (Part 2) (Active Comparator): Approximately 50 subjects will receive Carfilzomib 20 mg/m^2: Cycle 1, Day 1, 2. Carfilzomib 27 mg/m^2 (increased dosage of 27 mg/m^2 will be administered only if tolerated): Cycle 1, Days 8, 9 15, and 16; Cycle 2, Days 1, 2, 8, 9, 15 and 16 of each cycle; Cycle 3 and onwards, Days 1, 2, 8, 9, 15 and 16 of each cycle.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Afuresertib — Afuresertib will be dosed orally in morning, and will be sourced as opaque, white, size 4, 25 mg capsule and size 1, 100 mg capsules.
  Arms: Afuresertib 100 mg+ Carfilzomib (Part 1); Afuresertib 125 mg+ Carfilzomib (Part 1); Afuresertib 150 mg+ Carfilzomib (Part 1); Afuresertib/carfilzomib (Part 2)
Drug: Carfilzomib — Intravenous (IV) Carfilzomib will be sourced in the US from commercial stock. It will be a single-use 60 mg vial as a sterile, white to off-white lyophilized cake or powder

SUMMARY:
This open-label, 2-part Phase I/ randomized Phase II multi-center study is conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and clinical activity of afuresertib in combination with carfilzomib versus carfilzomib alone, in subjects with relapsed/refractory MM. Part 1 will evaluate 2 dose levels (125 milligrams [mg] and 150 mg of afuresertib) in 16 subjects (approximately 8 in each parallel arm) to determine an optimal dose of afuresertib for administration in combination with carfilzomib in Part 2. If neither of these dose levels are tolerated, an additional dose level of 100mg of afursertib in combination with carfilzomib may be explored in approximately 8 additional subjects. Part 2 was to investigate the safety, and clinical activity of the combination of afuresertib with carfilzomib (determined in Part 1) compared to carfilzomib alone, in approximately 100 subjects (50 in each parallel arm), however the study was terminated after the discontinuation of the single subject following the transition of the afuresertib development program from GSK to Novartis. The reason for the study termination is that the protocol defined study treatment was no longer aligned with the evolving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Histologically confirmed diagnosis of MM
* Received at least two prior therapies including bortezomib and an immunomodulatory agent and demonstrated disease progression on or within 60 days of completion of the last therapy. Subjects in Part 2 must also have measurable disease defined as having at least one of the following: Serum M-protein >=0.5 gram/ deciliter (g/dL) (>=5 gram/Liter [g/L]), Urine M-protein >=200 mg/24 hour (h), Serum free light chain (FLC) assay: Involved FLC level >=10 mg/dL (>=100 mg/L) and an abnormal serum free light chain ratio (<0.26 or >1.65), Biopsy proven plasmacytoma (should be measured within 28 days of the Screening Visit)
* Male or female, 18 years or older
* Performance status score of 0 - 1 according to the Eastern Cooperative Oncology Group (ECOG) scale
* Able to swallow and retain orally administered study treatment and does not have any clinically significant Gastro-intestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels or predispose subject to GI ulceration
* For the Alternate Arm (100 mg) only (if opened), willingness to undergo paired pre-dose and post-dose bone marrow aspirate and biopsies
* Fasting serum glucose <126 mg/dL (<7 millimole/liter [mmol/L]). Subjects diagnosed previously with Type 2 diabetes must also meet the additional following criteria: Controlled diabetes for >=6 months prior to enrolment, Hemoglobin A1c (HbA1c) =<8% at Screening visit
* Adequate organ system function defined as: Hematologic: Absolute neutrophil count (ANC) >=1.0 X 10/meter (m)^9/L, Hemoglobin >=8.0 g/dL, Platelets >=50 X 10 m^9/L, Prothrombin time/ International normalization ratio (PT/INR) <=1.5; Hepatic: Total bilirubin =<1.5 X Upper limit of normal (ULN) (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) =<1.5 X ULN, Serum Calcium corrected for albumin: =<12 mg/mL (=3 mmol/L); Cardiac: Corrected QT interval duration (QTc) interval <470 milliseconds (msecs), Left Ventricular Ejection Fraction (LVEF) (Echocardiogram [ECHO] or Multigated acquisition scan [MUGA]) >=50%, Renal: Serum Creatinine <2.5 mg/dL, Estimated glomerular filtration rate (GFR) or 24-hr urine creatinine clearance >=30 mL/ minute [min] (Estimated glomerular filtration rate will be calculated by the Modification of Diet in Renal Disease [MDRD] equation. When both a calculated and 24-hr creatinine clearance are available, the 24-hr value will be used). Note: Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may opt to retest the subject and the subsequent within range screening result may be used to confirm eligibility
* A female subject is eligible to participate if she is of Non-childbearing potential. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods as explained by the Investigator/designee, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. Child-bearing potential, has a negative serum pregnancy test within 7 days prior to start of study drugs, during the screening period, and agrees to use one of the contraception methods explained by the Investigator/designee from screening until four weeks after the last dose of afuresertib or carfilzomib
* Male subjects with female partners of child-bearing potential must have had a prior vasectomy or agree to use one of the contraception explained by the Investigator/designee. This criterion must be followed from the time of the first dose of study drugs until 10 days after the last dose of afuresertib or carfilzomib

Exclusion Criteria: Subjects meeting any of the following criteria must not be enrolled in the study:

* Prior treatment with carfilzomib and/or participation in any Phase 3 carfilzomib trial
* Chemotherapy, radiotherapy, immunotherapy, or other anti-myeloma therapy within 14 days prior to the first dose of any one of the drugs in the combination regimen. In addition, any drug-related toxicity should have recovered to Grade 1 or less
* Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of any one of the drugs in the combination regimen
* History of an allogeneic stem cell transplant
* Current use of prohibited medication during treatment with afuresertib
* Current chronic use of oral corticosteroids, with the exception of inhaled or topical steroids
* Unwillingness to follow the lifestyle and dietary restrictions
* Evidence of mucosal or internal bleeding
* Unresolved toxicity >=Grade 1 National Cancer Institute Common Terminology Criteria for Adverse Events, version 4 (NCI-CTCAE, 2009) from previous anti-cancer therapy except alopecia and <=Grade 2 peripheral neuropathy
* Any major surgery within the last four weeks
* Type 1 diabetes mellitus
* Any serious or unstable pre-existing medical, psychiatric disorder, or other condition (including lab abnormalities) that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following: Class II, III, or IV heart failure as defined by the New York Heart Association functional classification system; uncontrolled angina; clinically significant pericardial disease; severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant. Other clinically significant ECG abnormalities including second degree (Type II) or 3rd degree atrioventricular (AV) block; history of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening; pulmonary hypertension
* Known active infection requiring parenteral or oral anti-biotic treatment
* Previous or concurrent malignancies are allowed if it is clear that the other tumor is not contributing to the subject's illness. The subject must not be receiving active therapy, other than hormonal therapy, for this disease and the disease must be considered medically stable for at least 2 years.
* Pregnant or lactating female
* Known Human Immunodeficiency Virus (HIV) infection
* Subjects who are Hepatitis B surface antigen (HbSAg) positive. Subjects with a positive test for Hepatitis C (HCV) antibody are excluded, regardless of viral load. If hepatitis C antibody is positive, a confirmatory recombinant immunoblot assay (RIBA) test may be performed. If the RIBA test is negative, the subject is eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Part1: Number of participants with adverse events (AEs) as a measure of safety | Until 4 weeks after the last subject's last dose (LSLD) (Approximately assessed up to 4 years)
  AEs and serious adverse events (SAEs) will be collected from the screening until the follow-up visit
Part1: Safety assessed by monitoring the changes in vital signs | Until 4 weeks after the LSLD (Approximately assessed up to 4 years)
  Vital signs assessments included temperature, systolic and diastolic blood pressure, temperature and pulse rate measurements
Part1: Safety assessed by monitoring the changes in laboratory parameters | Until 4 weeks after the LSLD (Approximately assessed up to 4 years)
  Clinical laboratory parameters will include hematology and clinical chemistry
Part1: Safety assessed by monitoring the changes in electrocardiograms (ECG) | Until 4 weeks after the LSLD (Approximately assessed up to 4 years)
  Single 12-lead ECGs will be obtained over a brief recording period at the start of each cycle
Part 2: Progression Free Survivial (PFS) | Until 12 months of follow-up after the LSLD (Approximately assessed up to 6 years)
  PFS defined as the interval between the date of randomization and the earliest date of disease progression as assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Part 1: Composite of PK parameters of afuresertib and carfilzomib alone or in combination with each other will be assessed following multiple afuresertib doses and following a single dose of carfilzomib | Afuresertib (Cycle 1[C1], any Day[D] between 21-28 and C2 D1): 30 min predose; Carfilzomib (C1 D1 and C2 D1): 30 min predose; end of dosing; post dosing time-points for both treatments: 5 min, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12, 14-22, 24 hours (hr)
  Peripheral blood will be collected to evaluate PK parameters for Afuresertib (e.g., area under the plasma drug concentration-time curve [AUC], maximum observed plasma drug concentration [Cmax]) and carfilzomib (e.g., AUC, Cmax)
Part 1: Afuresertib concentrations | C1 D15: predose; 1 to 3 hr and 4 to 6 hr post-dose. C2 D1 and any cycle where disease assessments are obtained: pre-treatment and right before subject leaves clinic for the day (C2 and every 3rd cycle; approximately (approx) assessed up to 4 years)
  Afuresertib concentrations will be assessed in peripheral blood using a sparse sampling strategy
Part1: Overall response rate (ORR) | Until 12 months of follow-up after the LSLD (Approximately assessed up to 6 years)
  ORR is defined as the percentage of subjects with a confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as assessed by investigator using the 2011 recommendations in the International Myeloma Workshop Consensus (IMWC) Panel 1
Part1: PFS | Until 12 months of follow-up after the LSLD (Approximately assessed up to 6 years
  PFS is defined as the interval between the date of first dose and the earliest date of disease progression as assessed by investigator or death due to any cause
Part1: Overall survival (OS) | Until 12 months of follow-up after the LSLD (Approximately assessed up to 8 years
  OS is defined as the time until death due to any cause. Subjects will be followed for up to a maximum of 12 months following the LSLD. Subjects who are alive at 12 months following the LSLD will be censored for OS
Part1: Duration of response (DOR) | Until 12 months of follow-up after the LSLD (Approximately assessed up to 6 years)
  DOR defined for those subjects that achieve ORR as the time from first documented evidence of sCR, CR, VGPR, or PR until first documented disease progression or death
Part 2: ORR | Until 12 months of follow-up after LSLD (Approximately assessed up to 6 years)
  ORR defined as the percentage of subjects with a confirmed sCR, CR, VGPR or PR, as assessed by investigator using the 2011 recommendations in the IMWC Panel 1
Part 2: OS | Until 12 months of follow-up after the LSLD (Approximately assessed up to 8 years
  OS is defined as the time until death due to any cause. Subjects will be followed for up to a maximum of 12 months following the LSLD. Subjects who are alive at 12 months following the LSLD will be censored for OS
Part 2: DOR | Until 12 months of follow-up after LSLD (Approximately assessed up to 6 years)
  DOR defined for those subjects that achieve ORR as the time from first documented evidence of sCR, CR, VGPR, or PR until first documented disease progression or death
Part 2: Number of participants with adverse events (AEs) as a measure of safety | Until 4 weeks after the LSLD (Approximately assessed up to 4 years
  AEs and SAEs will be collected from the screening until the follow-up visit
Part 2: Safety assessed by monitoring the changes in vital signs | Until 4 weeks after the LSLD (Approximately assessed up to 4 years
  Vital signs assessments included temperature, systolic and diastolic blood pressure, temperature and pulse rate measurements
Part 2: Safety assessed by monitoring the changes in laboratory parameters | Until 4 weeks after the LSLD (Approximately assessed up to 4 years
  Clinical laboratory parameters will include hematology and clinical chemistry
Part 2: Safety assessed by monitoring the changes in ECG | Until 4 weeks after the LSLD (Approximately assessed up to 4 years
  Single 12-lead ECGs will be obtained over a brief recording period at the start of each cycle.
Part 2: Afuresertib concentrations | C1 D1: predose; 1-3 hr post-dose. C1 D15: predose; 1-3 hr and 4-6 hr post-dose. C2 D1 and any cycle where assessments are obtained: pre-treatment and right before subject leaves clinic for the day (C2 and every 3rd cycle; approx assessed up to 4 years)
  Afuresertib concentrations will be assessed in peripheral blood using a sparse sampling strategy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Cary, North Carolina, United States